CLINICAL TRIAL: NCT01099683
Title: A Double-blind, Randomised, Placebo-controlled Study in Elderly Subjects to Evaluate the Safety, Tolerability, Pharmacodynamic Effects and Pharmacokinetics of a Single Rectal Application of 10 mg NRL001 in a 2 g Suppository
Brief Title: Safety, Tolerability, Pharmacodynamic and Pharmacokinetics of a Single Rectal Application of 10 mg NRL001 in Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President Clinical Development, Norgine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NRL001-02/2009 (SAGE); 2009-017475-16 (EudraCT Number)
Record Dates: First submitted 2010-02-15; First posted 2010-04-07 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NRL001 (Experimental): All subjects will receive 10 mg NRL001 in a 2 g rectal suppository
  Interventions: Drug: NRL001
- Placebo (Placebo Comparator): All subjects will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NRL001 — Single rectal administration of 2 mg NRL001 in a 2 g suppository
  Arms: NRL001
Drug: Placebo — All subjects will receive rectal suppository containing placebo
  Arms: Placebo

SUMMARY:
A total of 26 healthy elderly male and female subjects will receive both 10 mg NRL001 in a 2 g rectal suppository and placebo in this double-blind, cross-over study. The order of treatment will be randomised, with a minimum washout period of 3 days between doses. An end of study assessment will be conducted at least 7 days after administration of the last treatment.

The pharmacokinetics of NRL001 will be determined prior to, and after, dosing. Pharmacodynamics will be examined using a three lead Holter monitor during both treatment periods. Adverse Events, vital signs, ECGs and clinical laboratory parameters will be collected, tabulated, reviewed and recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Volunteers will be included in the study if they satisfy the following criteria:

* Healthy adult male or female volunteers (as determined by medical history, physical examination, laboratory test values, vital signs and electrocardiograms [ECGs] at screening) aged ≥65 years.
* Non-smokers from 3 months before receiving the first dose and for the duration of the study.
* Body mass index (BMI) ≥ 18 and ≤ 32 kg/m2.
* Able and willing to receive rectal treatments.
* Able to voluntarily provide written informed consent to participate in the study.
* Sexually active male volunteers must use condoms with their partners throughout the study and for 90 days after completion of the study in addition to their partner's normal mode of contraception.
* Male volunteers must not donate sperm during the study and for 90 days after completion of the study.
* Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol.
* Female volunteers must be postmenopausal (for at least 1 year, confirmed by FSH testing at screening).
* Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).
* The volunteer's primary care physician must confirm that there is nothing in their medical history that would preclude their enrolment into this clinical study.

Exclusion Criteria:

Volunteers will be excluded if they fulfil any of the following criteria:

* Positive for HIV, hepatitis B, or hepatitis C as demonstrated by the results of testing at screening.
* History or presence of any significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal (GI), endocrine or immunologic disease.
* History or presence of any clinically significant ano-rectal conditions as judged by the Investigator (e.g. concomitant enlarged symptomatic haemorrhoids or acute presence of anal fissures) or clinically significant drug allergy.
* Blood pressure in excess of 150/90 mmHg or pulse rate below 50 beats per minute at screening.
* Any significant illness during the screening period preceding entry into this study.
* Clinically relevant ECG-abnormalities (e.g. QTc prolongation, acute arrhythmia) during the screening assessment
* Laboratory values which are abnormal and deemed to be clinically significant according to Bio-Kinetic Europe Ltd. SOPs, unless agreed in advance by the Sponsor's Responsible Medical Officer and the Bio-Kinetic Investigator.
* Current or history of drug or alcohol abuse or a positive drugs of abuse test at screening or check in.
* Use of any disallowed concomitant medication, including over-the-counter items within 14 days prior to study drug administration until the end of the study.
* Use of any medication applied via the rectum, within 30 days prior to dosing
* Use of any medication currently or within 30 days prior to dosing which the Investigator believes may affect the study participation or results.
* Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
* Donation of blood or blood products within 90 days prior to study drug administration, or at anytime during the study, except as required by this protocol.
* History of any allergy to medication, particularly nifedipine, α adrenoceptor antagonists or latex
* Consumption of alcoholic beverages within 24 hours prior to each dosing period. Abstinence is required during study confinement.
* Consumption of xanthine-containing products within 24 hours of each dosing period and during study confinement.
* Subjects who are considered not competent to consent to the trial or fail a Mini Mental State Exam (MMSE).
* Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic effects of NRL001 | 4 hours post-administration

SECONDARY OUTCOMES:
Pharmacokinetics of NRL001 | 30 hours post-administration
Safety will be assessed by recording adverse events (AEs), vital signs, 12-lead ECG, physical examinations and clinical laboratory tests. | Throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: David Bell, MRCGP MFPM, Principal Investigator — Bio-Kinetic Europe, Ltd.
Locations (1):
- Bio-Kinetic Europe Ltd, Belfast, United Kingdom

REFERENCES:
- [Derived] Bell D, Duffin A, Gruss HJ, Pediconi C, Jacobs A. A randomised, controlled, crossover study to investigate the pharmacodynamics, pharmacokinetics and safety of 1R,2S-methoxamine hydrochloride (NRL001) in healthy elderly subjects. Colorectal Dis. 2014 Mar;16 Suppl 1:27-35. doi: 10.1111/codi.12543. PMID 24499494